CLINICAL TRIAL: NCT06243575
Title: Comparison of Outcomes Between Multimodal Intraosseous Femoral Injection and Multimodal Intraosseous Tibial Injection, a Randomized Controlled Trial in Simultaneous Bilateral Total Knee Arthroplasty Patients
Brief Title: Comparison of Outcomes Between Intraosseous Femoral and Tibial Injection in Simultaneous Bilateral Total Knee Arthroplasty Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 149/66
Record Dates: First submitted 2024-01-16; First posted 2024-02-06 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-01

CONDITIONS: Pain, Postoperative
Keywords: total knee arthroplasty; intraosseous infiltration
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multimodal Intraosseous Femoral Injection (Experimental): Intraosseous injection of Ketorolac 15mg and Tranexamic acid 500mg in femoral canal
  Interventions: Drug: Multimodal Intraosseous Femoral Injection
- Multimodal Intraosseous Tibial Injection (Experimental): Intraosseous injection of Ketorolac 15mg and Tranexamic acid 500mg in tibial canal
  Interventions: Drug: Multimodal Intraosseous Tibial Injection

INTERVENTIONS:
Drug: Multimodal Intraosseous Femoral Injection — Intraosseous injection of Ketorolac 15mg and Tranexamic acid 500mg in femoral canal
  Arms: Multimodal Intraosseous Femoral Injection
Drug: Multimodal Intraosseous Tibial Injection — Intraosseous injection of Ketorolac 15mg and Tranexamic acid 500mg in tibial canal
  Arms: Multimodal Intraosseous Tibial Injection

SUMMARY:
In patients with osteoarthritis of the knee whose pain cannot be relieved by conservative treatment, total knee arthroplasty (TKA) is the operation that increases the quality of life for the patient. Pain management after total knee arthroplasty TKA is an important consideration to improve patient outcomes and reduce length of stay. Periarticular injections of the knee are one of the techniques used to reduce pain after surgery. Studies have shown that compared to other methods of pain relief, they are effective and safe. At present, no studies to compare between multimodal intraosseous femoral injection & multimodal intraosseous tibial injection in Simultaneous Bilateral TKA patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo bilateral Total knee Replacement due to osteoarthritis of both knees
* Used of a cemented, PS design TKA surgery.
* Able to give informed consent

Exclusion Criteria:

* Revision TKA
* History of previous knee or hip surgery
* History of allergic reaction or side effects to the drug that will be used in the experiment
* Underlying diseases of chronic kidney disease or chronic liver disease (Child Pugh B or C)
* Pregnancy
* History of coagulopathy or abnormal blood coagulation profile(INR >1.4 or aPTT ratio > 1.4)
* History of platelet dysfunction or platelet count < 140,0000/mm3
* History of Thromboembolism
* Use of Anticoagulants.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain score (Visual analog scale) | at 12 hours, 24 hours, 48 hours and 2 weeks after surgery
  Visual analog scale (VAS) score from 0-10(0 was no pain, 10 was worst pain ) between multimodal intraosseous femoral injection & multimodal intraosseous tibial injection

SECONDARY OUTCOMES:
Amount of painkillers used | up to 24 hours after surgery
Post operative blood loss | intraoperative and up to 48 hours postoperatively (include intraoperative and drain)
Knee and Osteoarthritis Outcome Score (KOOS) | post operative 2 weeks
  minimum and maximum values(0-100), higher scores mean a better outcome.
knee range of motion | post operative 2 weeks
Side effects and complications | intraoperative to post operative 2weeks
Length of hospital stay | Admit to discharge date (up to 7 days)
  Length of hospital stay record in number of days

CONTACTS AND LOCATIONS:
Overall Officials: Thakrit Chompoosang, MD, Study Director — Department of Medical Services Ministry of Public Health of Thailand
Locations (1):
- Rajavithi hospital, Phaya Thai, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brozovich AA, Incavo SJ, Lambert BS, Sullivan TC, Wininger AE, Clyburn TA, Taraballi F, Park KJ. Intraosseous Morphine Decreases Postoperative Pain and Pain Medication Use in Total Knee Arthroplasty: A Double-Blind, Randomized Controlled Trial. J Arthroplasty. 2022 Jun;37(6S):S139-S146. doi: 10.1016/j.arth.2021.10.009. Epub 2022 Mar 7. PMID 35272897
- [Background] Fan L, Zhu C, Zan P, Yu X, Liu J, Sun Q, Li G. The Comparison of Local Infiltration Analgesia with Peripheral Nerve Block following Total Knee Arthroplasty (TKA): A Systematic Review with Meta-Analysis. J Arthroplasty. 2015 Sep;30(9):1664-71. doi: 10.1016/j.arth.2015.04.006. Epub 2015 Apr 8. PMID 25922311